CLINICAL TRIAL: NCT03424265
Title: Effects of 12 Weeks of Nutritional Therapy Interventions in Heart Failure
Brief Title: Nutritional Therapy Interventions in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 206313
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure NYHA Class II
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9g of EAA mixture supplement (Experimental): Twice a day for 12 consecutive weeks.
  Interventions: Dietary Supplement: EAA mixture
- 9g of placebo (whey protein) (Experimental): Twice a day for 12 consecutive weeks.
  Interventions: Dietary Supplement: Placebo (whey protein)

INTERVENTIONS:
Dietary Supplement: EAA mixture — Dietary supplement intervention for 12-weeks
  Other Names: Essential Blends, Fairbanks, Alaska
  Arms: 9g of EAA mixture supplement
Dietary Supplement: Placebo (whey protein) — Dietary supplement intervention for 12-weeks
  Other Names: Pure Protein, 100% Whey Protein Powder, Bayport, NY
  Arms: 9g of placebo (whey protein)

SUMMARY:
The investigators will examine the effects of 12-weeks of nutritional interventions in older participants who have a symptom of mild to moderate heart failure.

DETAILED DESCRIPTION:
Heart failure develops when cardiac muscle becomes weakened and consequently is compromised in its ability to contract, relax, or both. Impaired heart function leads to reduced exercise capacity, which in turn leads to progressive muscle weakness and a vicious cycle of sedentary behavior, weight gain, and subsequent development of metabolic abnormalities and sarcopenia. Approximately 6-10% of individuals over the age of 65 suffer from heart failure, and the risk of death is 35% in the first year after diagnosis. In addition, there is a wide range of potential causes of heart failure, including the natural process of aging. Regardless of the specific underlying cause, there are common pathophysiological responses such as impaired exercise capacity, shortness of breath, fatigue and muscle strength, leading to decreased physical function. Moreover, some long-term consequences of reduced exercise tolerance and malabsorption in long-standing heart failure are loss of muscle mass and the development of cardiac cachexia, resulted in progression of sarcopenia. As protein and amino acid supplements are known to prevent loss of muscle mass or maintain muscle mass in alder individuals, in a pilot study 18 overweight/obese subjects with heart failure (all exceeded 40% body fat) were studied. Nine subjects received 12 weeks of dietary supplementation with 20 g of whey protein consumed daily, while the other nine were controls. The findings showed that supplementation with whey protein failed to improve functional performance as well as a limited stimulation of muscle protein synthesis. The lack of a demonstrable effect of whey protein is consistent with the diminished responsiveness to the stimulation of muscle protein synthesis. In contrast, a 2016 University of Arkansas for Medical Sciences (UAMS) pilot study found that the essential amino acid (EAA) mixture is better at overcoming anabolic resistance than Ensure Heart Health. In this study we will perform a randomized clinical trial of a commercially produced nutritional supplement as compared to a placebo in order to determine effects on physical function and health-related quality of life. Subjects will ingest either the EAA mixture product or placebo every day for 12 consecutive weeks. Outcomes will be determined by comparing the results of physical and functional tests from weeks -1 to 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 40 kg/m2
* Any ethnicity
* Presence of mild-to-moderate heart failure (NYHA II or III symptomatology) as evidenced by prescribed diuretics or reported shortness of breath upon exertion

Exclusion Criteria:

* Allergic to milk or soy products
* Hemoglobin <10 g/dL
* Estimated Glomerular Filtration Rate (eGFR) < 30
* Inability to perform strength and/or functional assessments
* Myocardial infarction in the past 6 months
* Unstable angina
* Moderate-severe heart valve disease
* Atrial fibrillation or other significant (as determined by PI) arrhythmias
* Infiltrative, restrictive or hypertrophic cardiomyopathy
* Dementia -determined by a SLUMS score of <20
* Currently having inflammatory bowel disease
* Received chemotherapy or radiation therapy within the past 12 months
* Currently undergoing tube feeding
* Currently receiving palliative care for end-of-life circumstance
* Unwilling to refrain from using non-study protein/amino acid supplements during their participation in this study
* If deemed medically unstable by the study physician for any other reason.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gohar Azhar, M.D, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azhar G, Verma A, Zhang X, Pangle A, Patyal P, Zhang W, Che Y, Coker K, Wolfe RR, Wei JY. Differential plasma protein expression after ingestion of essential amino acid-based dietary supplement verses whey protein in low physical functioning older adults. Geroscience. 2023 Jun;45(3):1729-1743. doi: 10.1007/s11357-023-00725-5. Epub 2023 Feb 1. PMID 36720768
- [Derived] Azhar G, Wei JY, Schutzler SE, Coker K, Gibson RV, Kirby MF, Ferrando AA, Wolfe RR. Daily Consumption of a Specially Formulated Essential Amino Acid-Based Dietary Supplement Improves Physical Performance in Older Adults With Low Physical Functioning. J Gerontol A Biol Sci Med Sci. 2021 Jun 14;76(7):1184-1191. doi: 10.1093/gerona/glab019. PMID 33475727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 9g of EAA Mixture Supplement | 9g of Placebo (Whey Protein)
Started | 29 | 34
Completed | 28 | 32
Not Completed | 1 | 2
Not completed — screening failure | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9g of EAA Mixture Supplement | 9g of Placebo (Whey Protein) | Total
Number analyzed (Participants) | 29 | 34 | 63
Age, Customized [Count of Participants; unit: Participants]
  Age >=60 years. | 29 | 34 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 25 | 28 | 53
  Asian | 1 | 0 | 1
  African-American | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Functional Test
Description: Measuring 6 minutes walking before and after the intervention. ***The results below are the actual increases of walking distance (mean and SD) changes from baseline to end of 12-week intervention.
Time Frame: Change from baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | 9g of EAA Mixture Supplement | 9g of Placebo (Whey Protein)
Number analyzed (Participants) | 28 | 32
feet | 115.91 (94.727) | 57.25 (150.527)

ADVERSE EVENTS:
Time Frame: Subjects were followed for adverse events for the duration of their participation (approx. 4 months).
Arm/Group | 9g of EAA Mixture Supplement | 9g of Placebo (Whey Protein)
All-Cause Mortality (participants affected / at risk) | 0/29 | 3/34
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/34
Other Adverse Events (participants affected / at risk) | 0/29 | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9g of EAA Mixture Supplement (N=29) | 9g of Placebo (Whey Protein) (N=34)
Prostate pain during urination (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory issue (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT03424265/Prot_SAP_000.pdf